CLINICAL TRIAL: NCT01789008
Title: Interest of Transient Elastography in the Determination of Advanced Fibrosis in Alcoholic Liver Didease in Alcoholic Patients in Weaning.
Brief Title: Transient Elastography in the Determination of Advanced Fibrosis in Alcoholic Liver Disease.
Acronym: FIBR-OH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PHRC/12-01; 2012-A01171-42
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2023-05-22 (Actual); Status verified 2018-09

CONDITIONS: Alcoholism; Liver Disease; Liver Fibrosis
Keywords: Transient elastography; Alcoholic liver disease; liver fibrosis
MeSH Terms: conditions — Alcoholism; Liver Diseases; Liver Cirrhosis; Liver Diseases, Alcoholic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transient elastography (Other): evaluation of fibrosis stage by transient elastography
  Interventions: Other: Determination of Advanced Fibrosis in Alcoholic Liver Disease
- liver biopsie (Active Comparator): evaluation of fibrosis stage by liver biopsie
  Interventions: Other: Determination of Advanced Fibrosis in Alcoholic Liver Disease

INTERVENTIONS:
Other: Determination of Advanced Fibrosis in Alcoholic Liver Disease

SUMMARY:
Alcoholic liver disease is the most frequent complication of excessive alcohol consumption. Early diagnosis of alcoholic liver disease is essential to avoid its complications that could be fatal. To date, the reference diagnostic tool is an invasive procedure: the liver biopsy. The transient elastography is a useful tool for early diagnosis of liver fibrosis. This tool is validated in the diagnosis of liver fibrosis due to C chronic hepatitis. Because it is non-invasive, fast, given immediate results; transient elastography could be repeated in alcoholic patients for liver fibrosis follow-up. In the present study, the investigators propose to realize liver biopsy and transient elastography in 300 alcoholic patients in weaning to evaluate the transient elastography accuracy in the exclusion of sever liver fibrosis (Metavir 3 and 4). The reference liver fibrosis diagnosis tool will be the liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years old; hospitalised for alcoholic weaning; with an alcoholic liver disease; with at risk alcoholic consumption; with an indication of liver biopsy; with a signed consentment.

Exclusion Criteria:

* patients with a cirrhosis; with other causes of liver disease; with a contraindication of liver biopsy; having had a liver biopsy in the last 3 years; pregnancy; major benefiting from a legal protective measure; no coverage care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Accuracy of transient elastography will be evaluated by AUC | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes university hospital, Rennes, France

REFERENCES:
- [Background] Chalin A, Turlin B, Ousmen A, Michalak S, Mueller J, Mueller S, Legros L, Bardou-Jacquet E, Viel JF, Samson M, Moirand R. Non-invasive diagnosis of alcohol-related steatohepatitis in patients ongoing alcohol withdrawal based on cytokeratin 18 and transient elastography. Aliment Pharmacol Ther. 2023 Jul;58(1):80-88. doi: 10.1111/apt.17515. Epub 2023 Apr 20. PMID 37078366
- [Result] Kiani A, Brun V, Laine F, Turlin B, Morcet J, Michalak S, Le Gruyer A, Legros L, Bardou-Jacquet E, Gandon Y, Moirand R. Acoustic radiation force impulse imaging for assessing liver fibrosis in alcoholic liver disease. World J Gastroenterol. 2016 May 28;22(20):4926-35. doi: 10.3748/wjg.v22.i20.4926. PMID 27239119
- [Derived] Legros L, Bardou-Jacquet E, Turlin B, Michalak S, Hamonic S, Le Gruyer A, Aziz K, Lemoine C, Bouvard N, Chavagnat JJ, Silvain C, Kerjean J, Le Dreau G, Lacave-Oberti N, Oberti F, Le Lan C, Guyader D, Moirand R. Transient Elastography Accurately Screens for Compensated Advanced Chronic Liver Disease in Patients With Ongoing or Recent Alcohol Withdrawal. Clin Gastroenterol Hepatol. 2022 Jul;20(7):1542-1552.e6. doi: 10.1016/j.cgh.2021.02.021. Epub 2021 Feb 12. PMID 33588101